CLINICAL TRIAL: NCT05642741
Title: Validation of a Self-questionnaire to Assess the Severity of Clinical Symptoms Related to Post-thyroidectomy Hypoparathyroidism
Brief Title: Validation of a Hypoparathyroidism Self-questionnaire
Acronym: SEV-HYPOPARA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Fondation SantéDige (Unknown); Association Francophone de Chirurgie Endocrinienne (AFCE) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC22_0495
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Thyroidectomy; Hypoparathyroidism Postprocedural
Keywords: Total thyroidectomy; Hypoparathyroidism Postprocedural; Quality of life; Self-questionnaire

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypoparathyroidism after total thyroidectomy: Adult patients definitive post-thyroidectomy HoPT defined by a parathyroid hormone (PTH) concentration ≤ 25 pg/mL more than 6 months after the operation and who require treatment with vitamin D and/or calcium supplementation. Each patient will complete a questionnaire twice (3 weeks apart +/- 7 days). The questionnaire, which evaluates the severity of clinical symptoms related to HoPT and their impact on quality of life, is adapted to this pathology.
  Interventions: Other: Response to medical and research questionnaires

INTERVENTIONS:
Other: Response to medical and research questionnaires — Patients will receive by mail or email the study information note, the medical questionnaire, the SF36 and the research questionnaire to be completed (then again 3 weeks later). The patients will return the questionnaires by mail or by post.

SUMMARY:
The aim of this study is to evaluate, for patients with post-thyroidectomy hypoparathyroidism (HoPT), the severity of their HoPT and to validate clinical scores from a self-administered questionnaire related to this disease (questionnaire which evaluates the severity of clinical symptoms related to HoPT and their impact on quality of life) in order to assess the severity of HoPT and to optimize support.

DETAILED DESCRIPTION:
Total thyroidectomy is a procedure very frequently performed in France (and worldwide. Around 35,000 patients are operated on each year in France. Among its complications, hypoparathyroidism (HoPT) results from a suppression or a significant decrease of parathyroid hormone (PTH) secretion leading to hypocalcemia associated with urinary calcium leakage.

The frequency of definitive HoPT (at least 6 months postoperative) varies from 1 to 10% (Sitges-Serra et al. Br J Surg, 2010, Duclos BMJ 2012). It is often underestimated by operators (Cho et al. Endocr Pract, 2014). Our team has previously shown that this HoPT is responsible for a significant impairment in quality of life (mental and physical) and voice (Frey et al. Ann Surg, 2021).

Despite the existence of treatment guidelines, only 26 to 32% of patients in French series are treated according to international recommendations (Bertocchio et al. Endocr Connect, 2022). It is therefore important to be able to assess the severity of HoPT and to validate a clinical score using a self-administered questionnaire related to this disease (questionnaire which assesses the severity of the clinical symptoms linked to HoPT and their impact on the quality of life).

Only patients with post-thyroidectomy HoPT will be included in the present study. Patients who underwent total thyroidectomy in the department of Loire-Atlantique will be prospectively included if they display post-operative HoPT. In addition, HoPT patients previously operated on and followed up in Loire-Atlantique, as well as patients from the "Hypoparathyroidisme France" association (https://hypopara.fr) and HoPT patients who have been included in the ThyrQol and Fothyr studies (Mirallié et al. Eur J Endocrinol, 2020, Blanchard et al. BJS Open, 2017) will also be included.The data collected will be routine biological data (usual blood and urine tests), responses to the SF36 questionnaire (validated quality of life questionnaire) and responses to a questionnaire that will assess the frequency and impact on the daily life of the symptoms reported by these patients. This questionnaire contains items related with symptoms that are frequently displayed by these patients and that are responsible for an impaired quality of life, in accordance with the data of the literature, our previous study (Frey et al. Ann Surg, 2021) and a discussion with the members of the association Hypoparathyroidism France.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patients undergoing total thyroidectomy
* Patients with permanent hypoparathyroidism defined by a parathyroid hormone concentration ≤ 25 pg/mL more than 6 months after surgery and who require vitamin and calcium therapy.
* Not being opposed to participating in the study (questionnaires will be sent with the study information note. If the patient returns the questionnaires: we will consider that he/she is not opposed to participate in this study)
* Participants must be affiliated to a social security system

Exclusion Criteria:

* Pregnant women when filling out questionnaires (the child's parathyroids can correct the mother's hypoparathyroidism)
* Minors or protected patients (under guardianship)
* Patients under court protection
* Patients on long-term vitamin-calcium therapy after total thyroidectomy whose PTH concentration has not been controlled or whose concentration is higher than 25 pg/mL.
* Hypoparathyroid patients of other origin than post-thyroidectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients who have undergone total thyroidectomy and who have definitive hypoparathyroidism
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Validate two clinical scores (a symptom importance score and a symptom impact score in daily life) from a questionnaire adapted to hypoparathyroidism, in order to better assess the severity of HoPT and optimize management. | 3 weeks
  To psychometrically validate the two scores created with the hypoparathyroidism severity questionnaire by showing, on the one hand, a good fit to a confirmatory two-dimensional factorial model (RSMEA<0.08 and CFI>0.9) and, on the other hand, by showing the good internal consistency of each of the scores (Cronbach's alpha >0.7).

SECONDARY OUTCOMES:
Discriminant validation : correlate hypoparathyroidism severity scores with biological results (PTH, calcemia, calciuria) | 3 weeks
  Discriminant validation: Spearman correlation coefficients between hypoparathyroidism severity questionnaire scores and biological results. Moderately strong values are expected (>0.4 in absolute value)
Concurrent validation of scores: correlate hypoparathyroidism severity scores with patients' quality of life scores (SF36) | 3 weeks
  Concurrent validation: Spearman correlation coefficients between hypoparathyroidism severity scores and SF36 quality of life scores. Negative correlations are expected (<-0.4)
Reproducibility of scores: show stability of scores at 3 week intervals (+/- 7 days) | 3 weeks
  Reproducibility: Intraclass correlation coefficients between the hypoparathyroidism severity scores obtained at two closely spaced questionnaire administrations (3 weeks apart +/- 1 week)

CONTACTS AND LOCATIONS:
Overall Officials: Eric MIRALLIE, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided